CLINICAL TRIAL: NCT05224141
Title: A Phase 3, Randomized, Double-Blind Study of MK-7684A in Combination With Etoposide and Platinum Followed by MK-7684A vs Atezolizumab in Combination With Etoposide and Platinum Followed by Atezolizumab for the First-Line Treatment of Participants With Extensive-Stage Small Cell Lung Cancer (KEYVIBE-008)
Brief Title: Pembrolizumab/Vibostolimab (MK-7684A) or Atezolizumab in Combination With Chemotherapy in First Line Treatment of Extensive-Stage Small Cell Lung Cancer (MK-7684A-008/KEYVIBE-008)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7684A-008; MK-7684A-008 (Other: MSD); KEYVIBE-008 (Other: MSD); jRCT2021220008 (Registry Identifier: jRCT); 2023-503517-30-00 (Registry Identifier: EU CT); U1111-1287-4436 (Registry Identifier: UTN); 2021-005034-42 (EudraCT Number)
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — pembrolizumab; Etoposide; Cisplatin; atezolizumab; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab/Vibostolimab (Experimental): Participants will receive 4 cycles (each cycle is 3 weeks) of a fixed-dose coformulation (FDC) of 200 mg pembrolizumab and 200 mg vibostolimab (MK-7684A) every 3 weeks (Q3W) via intravenous (IV) infusion, in combination with 100 mg/m^2 etoposide, and platinum (Area Under the Curve [AUC] 5 mg/mL/min carboplatin or 75 mg/m^2 cisplatin) chemotherapy Q3W for a total of approximately 12 weeks. This will be followed by additional cycles of MK-7684A (200 mg vibostolimab/200 mg pembrolizumab FDC) Q3W via IV infusion, until any of the conditions for discontinuation are met. To maintain the blinding, saline placebo will be administered on cycle 1 day 1 and then Q3W as needed beyond cycle 1.
  Interventions: Biological: Pembrolizumab/Vibostolimab Co-Formulation; Drug: Saline placebo; Drug: Etoposide; Drug: Cisplatin; Drug: Carboplatin
- Atezolizumab (Active Comparator): Participants will receive 4 cycles (each cycle is 3 weeks) of 1200 mg atezolizumab Q3W via IV infusion, in combination with 100 mg/m^2 etoposide and platinum (AUC 5 mg/mL/min carboplatin or 75 mg/m^2 cisplatin) chemotherapy Q3W for a total of approximately 12 weeks. This will be followed by additional cycles of atezolizumab (1200mg atezolizumab) Q3W via IV infusion until any of the conditions for discontinuation are met. To maintain the blinding, saline placebo will be administered on cycle 1 day 1 and then Q3W as needed beyond cycle 1.
  Interventions: Drug: Saline placebo; Drug: Etoposide; Drug: Cisplatin; Biological: Atezolizumab; Drug: Carboplatin

INTERVENTIONS:
Biological: Pembrolizumab/Vibostolimab Co-Formulation — Pembrolizumab 200 mg plus vibostolimab 200 mg fixed dose coformulation administered via IV infusion Q3W on Day 1 of each cycle until discontinuation criteria are met.
  Other Names: MK-7684A
  Arms: Pembrolizumab/Vibostolimab
Drug: Saline placebo — Saline solution administered via IV infusion on Cycle 1 (and Q3W as needed beyond Cycle 1)
Drug: Etoposide — Etoposide 100 mg/m^2 administered via IV infusion Q3W on Days 1 2, 3 of each cycle for up to 4 cycles
Drug: Cisplatin — Cisplatin 75 mg/m^2 administered via IV infusion Q3W on Day 1 of each cycle for up to 4 cycles.
  Other Names: PLATINOL-AQ®
Biological: Atezolizumab — Atezolizumab 1200 mg administered via IV infusion Q3W on Day 1 of each cycle until discontinuation criteria are met.
  Other Names: TECENTRIQ®
  Arms: Atezolizumab
Drug: Carboplatin — Carboplatin AUC 5 mg/mL/min administered via IV infusion Q3W on Day 1 of each cycle for up to 4 cycles.
  Other Names: PARAPLATIN®

SUMMARY:
This study will evaluate the combination of a fixed dose pembrolizumab/vibostolimab co-formulation (MK-7684A) with etoposide/platinum chemotherapy followed by MK-7684A compared to the combination of atezolizumab with etoposide/platinum chemotherapy followed by atezolizumab in the first-line treatment of Extensive-Stage Small Cell Lung Cancer (ES-SCLC). The primary hypothesis is, with respect to overall survival, MK-7684A in combination with the background therapy of etoposide/platinum followed by MK-7684A, is superior to atezolizumab in combination with the background therapy of etoposide/platinum followed by atezolizumab.

DETAILED DESCRIPTION:
With Amendment 4, the experimental Pembrolizumab/Vibostolimab arm (MK-7684A) was discontinued and all ongoing participants were offered an option to move to the comparator Atezolizumab monotherapy arm for the remainder of the study. There will be no further analyses of efficacy, and no European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire-Core 30 (QLQ-C30) and Lung Cancer 13 module (EORTC QLQ-LC13) outcome measures will be reported.

Effective as of Amendment 5, participants with access to approved standard of care (SOC) should be considered for discontinuation from the study. Those benefiting from atezolizumab, but unable to access it as SOC outside the study, may continue on study and receive treatment with atezolizumab until discontinuation criteria are met.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has histologically or cytologically confirmed diagnosis of extensive-stage small cell lung cancer (ES-SCLC) in need of first-line therapy
* Has ES-SCLC defined as Stage IV (T any, N any, M1a/b/c) by the American Joint Committee on Cancer, Eighth Edition or T3-T4 due to multiple lung nodules that are too extensive or have tumor/nodal volume that is too large to be encompassed in a tolerable radiation plan
* Males agree to use contraception, refrain from donating sperm, and abstain from heterosexual intercourse
* Females are not pregnant or breastfeeding, is not a woman of childbearing potential (WOCBP) or is a WOCBP who uses a highly effective contraceptive method, or is abstinent from heterosexual intercourse
* Has measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
* Has a predicted life expectancy of >3 months

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Is considered a poor medical risk due to a serious, uncontrolled medical disorder or non-malignant systemic disease
* Has received prior treatment for Small Cell Lung Cancer (SCLC)
* Is expected to require any other form of antineoplastic therapy for SCLC while on study
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has a history of severe hypersensitivity reaction (≥Grade 3) to any study intervention and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has a known history of, or active, neurologic paraneoplastic syndrome
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B or known active Hepatitis C virus infection
* Has had an allogenic tissue/solid organ transplant
* Has had major surgery within prior 3 weeks or has not recovered adequately from toxicity and/or complications from an intervention prior to receiving the first dose of study intervention
* Has symptomatic ascites or pleural effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2027-06-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (140):
- United States (11):
  - Infirmary Cancer Care ( Site 0022), Mobile, Alabama
  - Los Angeles Hematology Oncology Medical Group ( Site 0006), Los Angeles, California
  - VA West Los Angeles Medical Center ( Site 0004), Los Angeles, California
  - Boca Raton Regional Hospital-Lynn Cancer Institute ( Site 0014), Boca Raton, Florida
  - Fort Wayne Medical Oncology and Hematology ( Site 0013), Fort Wayne, Indiana
  - Dana-Farber Cancer Institute ( Site 0018), Boston, Massachusetts
  - Cancer and Hematology Centers of Western Michigan ( Site 0001), Grand Rapids, Michigan
  - Hattiesburg Clinic Hematology/Oncology ( Site 0003), Hattiesburg, Mississippi
  - Lancaster General Hospital - Ann B Barshinger Cancer Institute ( Site 0005), Lancaster, Pennsylvania
  - Blue Ridge Cancer Care ( Site 0015), Blacksburg, Virginia
  - University of Virginia Cancer Center ( Site 0019), Charlottesville, Virginia
- Argentina (5):
  - Hospital Italiano de Buenos Aires-Clinical Oncology ( Site 0203), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0201), Mar del Plata, Buenos Aires
  - Centro de Educación Médica e Investigaciones Clínicas (CEMIC)-Medical Oncology ( Site 0200), Buenos Aires, Buenos Aires F.D.
  - Hospital Provincial del Centenario ( Site 0205), Rosario, Santa Fe Province
  - Sanatorio Parque ( Site 0202), Rosario, Santa Fe Province
- Australia (4):
  - Nepean Hospital ( Site 2700), Kingswood, New South Wales
  - Calvary Mater Newcastle ( Site 2703), Waratah, New South Wales
  - Frankston Hospital-Oncology and Haematology ( Site 2702), Frankston, Victoria
  - Western Health-Sunshine & Footscray Hospitals-Cancer Services-Cancer Research ( Site 2701), Melbourne, Victoria
- Austria (5):
  - Medizinische Universität Graz ( Site 0504), Graz, Styria
  - Ordensklinikum Linz GmbH Elisabethinen-Department of Pneumology ( Site 0505), Linz, Upper Austria
  - Kepler Universitätsklinikum ( Site 0507), Linz, Upper Austria
  - Standort Penzing der Klinik Ottakring-Abteilung für Atemwegs-und Lungenkrankheiten ( Site 0502), Vienna
  - Klinik Floridsdorf-Abteilung für Innere Medizin und Pneumologie ( Site 0501), Vienna
- Canada (2):
  - Kingston Health Sciences Centre-Kingston General Hospital Site ( Site 0106), Kingston, Ontario
  - Lakeridge Health ( Site 0102), Oshawa, Ontario
- China (19):
  - Anhui Cancer Hospital ( Site 2915), Hefei, Anhui
  - Beijing Cancer hospital-Thoracic Cancer Department A ( Site 2901), Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital ( Site 2921), Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital-oncology department ( Site 2904), Fuzhou, Fujian
  - Harbin Medical University Cancer Hospital-oncology of department ( Site 2920), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 2916), Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology-Medical Oncology ( Site 2912), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 2922), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 2907), Changsha, Hunan
  - The First Affiliated Hospital of Soochow University ( Site 2913), Suzhou, Jiangsu
  - Jilin Cancer Hospital-GCP office ( Site 2909), Changchun, Jilin
  - The First Hospital of Jilin University ( Site 2914), Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University-Oncology ( Site 2910), Xi'an, Shaanxi
  - Shanghai Chest Hospital-Oncology department ( Site 2900), Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center ( Site 2908), Shanghai, Shanghai Municipality
  - Sichuan Cancer hospital. ( Site 2923), Chengdu, Sichuan
  - West China Hospital Sichuan University ( Site 2903), Chengdu, Sichuan
  - Sir Run Run Shaw Hospital-Medical Oncology ( Site 2906), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital-Oncology ( Site 2919), Hangzhou, Zhejiang
- Finland (3):
  - Oulun yliopistollinen sairaala-Oncology and Hematology ( Site 0702), Oulu, North Ostrobothnia
  - Vaasan Keskussairaala-Department of Clinical Oncology ( Site 0700), Vaasa, Pohjanmaa
  - Turku University Hospital-The Department of Pulmonary Medicine ( Site 0701), Turku, Southwest Finland
- France (3):
  - Assistance Publique Hôpitaux de Marseille - Hôpital Nord ( Site 0805), Marseille, Bouches-du-Rhone
  - CHU de Toulouse - Hopital Larrey-service de pneumologie ( Site 0800), Toulouse, Haute-Garonne
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuyt-Unité d'oncologie thoracique et cutané ( Site 0803), Limoges, Haute-Vienne
- Germany (5):
  - Thoraxklinik-Heidelberg gGmbH-Studienzentrum Thoraxonkologie ( Site 0905), Heidelberg, Baden-Wurttemberg
  - Lungenfachklinik Immenhausen-Thoracic Oncology ( Site 0907), Immenhausen, Hesse
  - Medizinische Hochschule Hannover-Department of Pneumology ( Site 0901), Hanover, Lower Saxony
  - LungenClinic Grosshansdorf-Onkologie ( Site 0903), Großhansdorf, Schleswig-Holstein
  - SRH Wald-Klinikum Gera-Lungenkrebszentrum ( Site 0900), Gera, Thuringia
- Greece (5):
  - Errikos Dunant Hospital Center-Second Department of Oncology and Clinical Trials Unit ( Site 1002), Athens, Attica
  - Sotiria Thoracic Diseases Hospital of Athens ( Site 1003), Athens, Attica
  - Metropolitan Hospital ( Site 1001), Athens, Attica
  - University General Hospital of Heraklion ( Site 1004), Heraklion, Irakleio
  - European Interbalkan Medical Center ( Site 1000), Thessaloniki
- Hungary (4):
  - Bacs-Kiskun Megyei Korhaz-Onkoradiologiai Kozpont ( Site 1105), Kecskemét, Bács-Kiskun county
  - Petz Aladar Egyetemi Oktato Korhaz-Pulmonológia (Dr. Szalai Zsuzsanna) ( Site 1102), Győr, Győr-Moson-Sopron
  - Reformatus Pulmonologiai Centrum-Onkopulmonologiai Jarobeteg Centrum ( Site 1101), Törökbálint, Pest County
  - Somogy Megyei Kaposi Mór Oktató Kórház-Pulmonologiai Osztaly ( Site 1104), Kaposvár, Somogy County
- Ireland (2):
  - St. James's Hospital ( Site 1200), Dublin
  - Beaumont Hospital, Dublin-Cancer Clinical Trials & Research Unit ( Site 1201), Dublin
- Israel (3):
  - Rambam Health Care Campus-Oncology ( Site 1301), Haifa
  - Shaare Zedek Medical Center-Oncology ( Site 1300), Jerusalem
  - Sheba Medical Center-ONCOLOGY ( Site 1302), Ramat Gan
- Italy (4):
  - Azienda Ospedaliera Dei Colli-U.O.C Pneumologia Oncologica DH PNL ONC ( Site 1402), Naples, Campania
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 1401), Milan, Lombardy
  - Humanitas-U.O di Oncologia medica ed Ematologia ( Site 1403), Rozzano, Milano
  - Istituto Nazionale Tumori Regina Elena-Oncologia Medica 2 ( Site 1400), Rome, Roma
- Japan (14):
  - Aichi Cancer Center ( Site 3016), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 3002), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 3012), Matsuyama, Ehime
  - Kurume University Hospital ( Site 3014), Kurume, Fukuoka
  - National Hospital Organization Hokkaido Cancer Center ( Site 3015), Sapporo, Hokkaido
  - Kanazawa University Hospital ( Site 3006), Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center ( Site 3004), Yokohama, Kanagawa
  - Sendai Kousei Hospital ( Site 3001), Sendai, Miyagi
  - Niigata Cancer Center Hospital ( Site 3005), Niigata, Niigata
  - Kansai Medical University Hospital ( Site 3009), Hirakata, Osaka
  - Shizuoka Cancer Center ( Site 3007), Nakatogari, Shizuoka
  - Cancer Institute Hospital of JFCR ( Site 3003), Koto, Tokyo
  - National Hospital Organization Kyushu Medical Center ( Site 3013), Fukuoka
  - Okayama University Hospital ( Site 3011), Okayama
- Lithuania (3):
  - Klaipeda University Hospital-Oncology chemotherapy ( Site 1502), Klaipėda, Klaipedos Miestas
  - National Cancer Institute-Department of Thoracic Surgery and Oncology ( Site 1501), Vilnius, Vilniaus Miestas
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos-Pulmonology ( Site 1500), Kaunas
- Mexico (5):
  - Hospital Civil Fray Antonio Alcalde-Oncology ( Site 0407), Guadalajara, Jalisco
  - Actualidad Basada en la Investigación del Cáncer-Lung Cancer ( Site 0403), Guadalajara, Jalisco
  - Arké SMO S.A. de C.V. ( Site 0401), Mexico City, Mexico City
  - iCan Oncology Center Centro Medico AVE ( Site 0406), Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca ( Site 0410), Oaxaca City
- Netherlands (7):
  - Ziekenhuis Rijnstate ( Site 1606), Arnhem, Gelderland
  - Maastricht UMC+-Pulmonary disease ( Site 1602), Maastricht, Limburg
  - Jeroen Bosch Hospital-Pulmonology ( Site 1605), 's-Hertogenbosch, North Brabant
  - Isala, locatie Zwolle-Poli Longziekten ( Site 1612), Zwolle, Overijssel
  - Medische Centrum Leeuwarden ( Site 1619), Leeuwarden, Provincie Friesland
  - Erasmus Medisch Centrum ( Site 1621), Rotterdam, South Holland
  - Martini Ziekenhuis ( Site 1618), Groningen
- Poland (7):
  - Przychodnia Lekarska KOMED ( Site 1701), Konin, Greater Poland Voivodeship
  - Med-Polonia Sp. z o. o. ( Site 1710), Poznan, Greater Poland Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 1709), Siedlce, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier ( Site 1700), Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 1703), Przemyśl, Podkarpackie Voivodeship
  - Szpital Specjalistyczny w Prabutach Spolka z o.o. ( Site 1706), Prabuty, Pomeranian Voivodeship
  - Centrum Pulmonologii i Torakochirurgii w Bystrej ( Site 1707), Bystra, Silesian Voivodeship
- Portugal (4):
  - Champalimaud Foundation ( Site 1812), Lisbon, Lisbon District
  - Hospital CUF Descobertas ( Site 1815), Lisbon, Lisbon District
  - Centro Hospitalar do Porto - Hospital de Santo António ( Site 1813), Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE ( Site 1810), Porto
- Romania (6):
  - MedEuropa Bucuresti - Centru de Radioterapie-Oncology ( Site 1905), Bucharest, București
  - Centrul medical Focus ( Site 1903), Bucharest, București
  - Cardiomed SRL Cluj-Napoca ( Site 1900), Cluj-Napoca, Cluj
  - Centrul de Oncologie Oncolab-Medical Oncology ( Site 1904), Craiova, Dolj
  - Centrul de Oncologie Sfantul Nectarie-Medical ( Site 1901), Craiova, Dolj
  - Cabinet Medical Oncomed ( Site 1902), Timișoara, Timiș County
- South Korea (4):
  - Chonnam National University Hwasun Hospital-Pulmonology ( Site 2800), Hwasun, Jeonranamdo
  - Kyungpook National University Chilgok Hospital-Pulmonology ( Site 2801), Deagu, Taegu-Kwangyokshi
  - Chungnam national university hospital-Department of Internal Medicine ( Site 2802), Daejeon, Taejon-Kwangyokshi
  - Korea University Guro Hospital-Internal Medicine ( Site 2803), Seoul
- Spain (4):
  - Hospital Universitario 12 de Octubre-Medical Oncology ( Site 2102), Madrid, Madrid, Comunidad de
  - H.R.U Málaga - Hospital General-Oncology ( Site 2104), Málaga, Malaga
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 2100), Barcelona
  - Hospital Universitario Virgen Macarena-Unidad de Investigación Oncológica ( Site 2103), Seville
- Turkey (Türkiye) (8):
  - Ege University Medicine of Faculty-Chest Diseases Department ( Site 2402), Bornova, İzmir
  - Baskent University Dr. Turgut Noyan Research and Training Center-ONCOLOGY ( Site 2407), Adana
  - Hacettepe Universitesi-oncology hospital ( Site 2409), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 2406), Ankara
  - Ankara Bilkent City Hospital ( Site 2403), Ankara
  - Medipol University Medical Faculty-oncology ( Site 2400), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 2401), Istanbul
  - I.E.U. Medical Point Hastanesi-Oncology ( Site 2408), Izmir
- United Kingdom (3):
  - The Christie-Clinical Research Facility ( Site 2607), Manchester, England
  - Mount Vernon Hospital ( Site 2602), Northwood, Hillingdon
  - Heartlands Hospital-Oncology Research ( Site 2604), Birmingham

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Shapira-Frommer R, Niu J, Perets R, Peters S, Shouse G, Lugowska I, Garassino MC, Sands J, Keenan T, Zhao B, Healy J, Ahn MJ. The KEYVIBE program: vibostolimab and pembrolizumab for the treatment of advanced malignancies. Future Oncol. 2024;20(27):1983-1991. doi: 10.1080/14796694.2024.2343272. Epub 2024 Sep 4. PMID 39230120
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26261&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab/Vibostolimab: Participants received 4 cycles (each cycle is 3 weeks) of a fixed-dose coformulation (FDC) of 200 mg pembrolizumab and 200 mg vibostolimab (MK-7684A) every 3 weeks (Q3W) via intravenous (IV) infusion, in combination with 100 mg/m^2 etoposide, and platinum (Area Under the Curve [AUC] 5 mg/mL/min carboplatin or 75 mg/m^2 cisplatin) chemotherapy Q3W for a total of approximately 12 weeks. This was followed by additional cycles of MK-7684A (200 mg vibostolimab/200 mg pembrolizumab FDC) Q3W via IV infusion, until any of the conditions for discontinuation are met. To maintain the blinding, saline placebo was administered on cycle 1 day 1 and then Q3W as needed beyond cycle 1.
- Atezolizumab: Participants received 4 cycles (each cycle is 3 weeks) of 1200 mg atezolizumab Q3W via IV infusion, in combination with 100 mg/m^2 etoposide and platinum (AUC 5 mg/mL/min carboplatin or 75 mg/m^2 cisplatin) chemotherapy Q3W for a total of approximately 12 weeks. This was followed by additional cycles of atezolizumab (1200mg atezolizumab) Q3W via IV infusion until any of the conditions for discontinuation are met. To maintain the blinding, saline placebo was administered on cycle 1 day 1 and then Q3W as needed beyond cycle 1.
Period: Overall Study
Arm/Group | Pembrolizumab/Vibostolimab | Atezolizumab
Started | 230 | 230
Treated | 229 | 229
Completed | 0 | 0
Not Completed | 230 | 230
Not completed — Ongoing | 75 | 88
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Death | 153 | 138

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab/Vibostolimab | Atezolizumab | Total
Number analyzed (Participants) | 230 | 230 | 460
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (8.8) | 63.9 (8.5) | 63.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 64 | 140
  Male | 154 | 166 | 320
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 18 | 30
  Not Hispanic or Latino | 213 | 209 | 422
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 78 | 64 | 142
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 135 | 158 | 293
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 10 | 4 | 14
Eastern Cooperative Oncology Group (ECOG) Performance Status at Baseline [Count of Participants; unit: Participants] — An ECOG Performance Status at baseline; ECOG= 0 (Fully active, able to carry on all pre-disease performance without restriction), or ECOG= 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature) was required for participant inclusion in the study and randomization was stratified by baseline ECOG score.
  Participants
    ECOG= 0 | 77 | 81 | 158
    ECOG= 1 | 153 | 149 | 302
Lactate Dehydrogenase (LDH) Status at Baseline [Count of Participants; unit: Participants] — Randomization of participants in the study was stratified by LDH measurement at baseline (≤ or > upper limit of normal [ULN]).
  Participants
    ≤Upper Limit of Normal (ULN) | 92 | 94 | 186
    >Upper Limit of Normal (ULN) | 138 | 136 | 274
Presence of Liver Metastases at Baseline [Count of Participants; unit: Participants] — Randomization of participants in the study was stratified by the presence of liver metastases at baseline (yes or no).
  Participants
    Yes | 93 | 98 | 191
    No | 137 | 132 | 269
Presence of Brain Metastases at Baseline [Count of Participants; unit: Participants] — Randomization of participants in the study was stratified by the presence of brain metastases at baseline (yes or no).
  Participants
    Yes | 15 | 15 | 30
    No | 215 | 215 | 430

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. OS was calculated using the nonparametric Kaplan-Meier method for censored data.
Time Frame: Up to approximately 25 months
Population: Per protocol, the analysis population consisted of all randomized participants who were included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab/Vibostolimab | Atezolizumab
Number analyzed (Participants) | 230 | 230
Months | 11.5 [9.8 to 12.6] | 12.9 [11.6 to 14.8]
Statistical Analysis 1: Comparison: Pembrolizumab/Vibostolimab vs Atezolizumab; Statistical analyses stratified by ECOG performance status (0 vs. 1), LDH (≤ULN vs. >ULN), liver metastasis (Yes or No), and brain metastasis (Yes or No); Test type: Superiority; p = 0.9762, Log Rank; One-sided p-value based on log-rank test stratified by ECOG performance status, LDH, liver metastasis, and brain metastasis; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [1.00 to 1.59] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG performance status (0 vs. 1), LDH (≤ULN vs. >ULN), liver metastasis (Yes or No), and brain metastasis (Yes or No)

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. Per protocol, RECIST 1.1 was modified to allow up to 10 target lesions total (up to 5 per organ). PFS was calculated using the nonparametric Kaplan-Meier method; participants who did not experience a PFS event were censored at the last disease assessment, or the last assessment before new anticancer treatment if new treatment was initiated. PFS as assessed by blinded independent central review (BICR) per RECIST 1.1 is presented.
Time Frame: Up to approximately 25 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab/Vibostolimab | Atezolizumab
Number analyzed (Participants) | 230 | 230
Months | 5.3 [4.4 to 5.4] | 4.5 [4.4 to 5.3]
Statistical Analysis 1: Comparison: Pembrolizumab/Vibostolimab vs Atezolizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5316, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.82 to 1.23] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants in the analysis population who have a confirmed Complete Response (CR: disappearance of all lesions) or a Partial Response (PR: ≥30% decrease in the sum of target lesion diameters without progression in other lesions) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR). Per protocol, RECIST 1.1 was modified to allow up to 10 target lesions total (up to 5 per organ). The ORR was calculated using the Miettinen & Nurminen method stratified by baseline ECOG performance status (0 or 1), baseline LDH (≤ or > upper limit of normal [ULN]), and baseline presence of liver metastasis (Yes or No), or brain metastasis (Yes or No).
Time Frame: Up to approximately 25 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab/Vibostolimab | Atezolizumab
Number analyzed (Participants) | 230 | 230
Percentage of Participants | 71.7 [65.4 to 77.5] | 74.8 [68.7 to 80.3]
Statistical Analysis 1: Comparison: Pembrolizumab/Vibostolimab vs Atezolizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Percent Difference = -3.1, 95% CI 2-sided [-11.1 to 4.9] — Based on Miettinen & Nurminen method stratified by ECOG performance status (0 vs. 1), LDH (≤ULN vs. >ULN), liver metastasis (Yes or No), and brain metastasis (Yes or No)

4. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrated a confirmed Complete Response (CR: disappearance of all lesions) or Partial Response (PR: ≥30% decrease in the sum of target lesion diameters without progression in other lesions) per RECIST 1.1, DOR was defined as the time from first documented CR or PR until progressive disease (PD) or death from any cause, whichever occurs first. Per protocol, RECIST 1.1 was modified to allow up to 10 target lesions total (up to 5 per organ). DOR was calculated using the nonparametric Kaplan-Meier method for censored data.
Time Frame: Up to approximately 25 months
Population: Per protocol, the analysis population consisted of all randomized participants who were included in the treatment group to which they were randomized and experienced a CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab/Vibostolimab | Atezolizumab
Number analyzed (Participants) | 165 | 172
Months | 4.2 [4.1 to 4.3] | 3.9 [3.4 to 4.1]

5. Secondary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to approximately 60 months
Reporting Status: Not Posted

6. Secondary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to an AE
Description: as for outcome 5
Time Frame: Up to approximately 60 months
Reporting Status: Not Posted

7. Secondary Outcome: Change From Baseline in the Global Health Status/Quality of Life (Items 29 and 30) Combined Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Description: The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life (QoL) of individuals with cancer. Participant responses to Items 29 and 30 ("How would you rate your overall health during the past week?" and "How would you rate your overall QoL during the past week?") are scored on a 7-point scale (1=Very Poor to 7=Excellent). A higher score indicates a better overall outcome.
Time Frame: Baseline and up to approximately 60 months
Reporting Status: Not Posted

8. Secondary Outcome: Change From Baseline in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30
Description: The EORTC QLQ-C30 is a cancer specific health-related QoL questionnaire. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a worse level of function.
Time Frame: Baseline and up to approximately 60 months
Reporting Status: Not Posted

9. Secondary Outcome: Change From Baseline in Dyspnea Score (Item 8) on the EORTC QLQ-C30
Description: The EORTC QLQ-C30 is a cancer specific health-related QoL questionnaire. Participant response to the question "Were you short of breath?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of dyspnea.
Time Frame: Baseline and up to approximately 60 months
Reporting Status: Not Posted

10. Secondary Outcome: Change From Baseline in Cough Score (Item 31) on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13)
Description: The EORTC QLQ-LC13 is a lung cancer specific health-related QoL questionnaire. Participant response to the question "Have you coughed?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates more frequent coughing.
Time Frame: Baseline and up to approximately 60 months
Reporting Status: Not Posted

11. Secondary Outcome: Change From Baseline in Chest Pain Score (Item 40) on the EORTC QLQ-LC13
Description: EORTC QLQ-LC13 is a lung cancer specific health-related QoL questionnaire. Participant response to the question "Have you had pain in your chest?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of chest pain.
Time Frame: Baseline and up to approximately 60 months
Reporting Status: Not Posted

12. Secondary Outcome: Time to True Deterioration (TTD) in the Global Health Status/Quality of Life (Items 29 and 30) Combined Score on the EORTC QLQ-C30
Description: The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the QoL of individuals with cancer. Participant responses to Items 29 and 30 ("How would you rate your overall health during the past week?" and "How would you rate your overall QoL during the past week?") are scored on a 7-point scale (1=Very Poor to 7=Excellent). A higher score indicates a better overall outcome. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Baseline and up to approximately 60 months
Reporting Status: Not Posted

13. Secondary Outcome: TTD in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30
Description: The EORTC QLQ-C30 is a cancer specific health-related QoL questionnaire. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a worse level of function. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Baseline and up to approximately 60 months
Reporting Status: Not Posted

14. Secondary Outcome: TTD in Dyspnea Score (Item 8) on the EORTC QLQ-C30
Description: The EORTC QLQ-C30 is a cancer specific health-related QoL questionnaire. Participant response to the question "Were you short of breath?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of dyspnea. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Baseline and up to approximately 60 months
Reporting Status: Not Posted

15. Secondary Outcome: TTD in Cough Score (Item 31) on the EORTC QLQ-LC13
Description: The EORTC QLQ-LC13 is a lung cancer specific health-related QoL questionnaire. Participant response to the question "Have you coughed?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates more frequent coughing. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Baseline and up to approximately 60 months
Reporting Status: Not Posted

16. Secondary Outcome: TTD in Chest Pain Score (Item 40) on the EORTC QLQ-LC13
Description: The EORTC QLQ-LC13 is a lung cancer specific health-related QoL questionnaire. Participant response to the question "Have you had pain in your chest?" is scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a worse level of chest pain. TTD is defined as the time to first onset of 10 or more (out of 100) deterioration from baseline and confirmed by a second adjacent 10 or more deterioration from baseline.
Time Frame: Baseline and up to approximately 60 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to approximately 25 months
Description: All-cause mortality was reported on all randomized participants. Serious and non-serious adverse events (AEs) were reported on all randomized participants who received ≥1 dose of treatment. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | Pembrolizumab/Vibostolimab | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 155/230 | 141/230
Serious Adverse Events (participants affected / at risk) | 120/229 | 96/229
Other Adverse Events (participants affected / at risk) | 228/229 | 222/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab/Vibostolimab (N=229) | Atezolizumab (N=229)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 8 (8)
Febrile neutropenia (Blood and lymphatic system disorders) | 15 (16) | 13 (13)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 7 (7)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Dilated cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 3 (3) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0)
Immune-mediated adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 6 (6) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0)
General physical health deterioration (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1)
Infusion related hypersensitivity reaction (Immune system disorders) | 1 (1) | 0 (0)
Amoebic dysentery (Infections and infestations) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 3 (3) | 0 (0)
Encephalitis cytomegalovirus (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 19 (20) | 17 (19)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Immune-mediated encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aneurysm ruptured (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava occlusion (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab/Vibostolimab (N=229) | Atezolizumab (N=229)
Anaemia (Blood and lymphatic system disorders) | 154 (228) | 130 (181)
Leukopenia (Blood and lymphatic system disorders) | 95 (259) | 87 (187)
Lymphopenia (Blood and lymphatic system disorders) | 25 (50) | 14 (28)
Neutropenia (Blood and lymphatic system disorders) | 130 (320) | 126 (260)
Thrombocytopenia (Blood and lymphatic system disorders) | 80 (157) | 73 (128)
Hyperthyroidism (Endocrine disorders) | 23 (24) | 23 (27)
Hypothyroidism (Endocrine disorders) | 38 (50) | 22 (26)
Abdominal pain upper (Gastrointestinal disorders) | 12 (14) | 8 (10)
Constipation (Gastrointestinal disorders) | 60 (76) | 68 (81)
Diarrhoea (Gastrointestinal disorders) | 45 (56) | 46 (59)
Nausea (Gastrointestinal disorders) | 85 (141) | 82 (134)
Vomiting (Gastrointestinal disorders) | 39 (55) | 19 (27)
Asthenia (General disorders) | 47 (59) | 40 (61)
Chest pain (General disorders) | 7 (8) | 13 (14)
Fatigue (General disorders) | 58 (72) | 51 (55)
Malaise (General disorders) | 13 (18) | 9 (14)
Oedema peripheral (General disorders) | 14 (14) | 11 (11)
Pyrexia (General disorders) | 24 (25) | 23 (24)
COVID-19 (Infections and infestations) | 32 (34) | 35 (37)
Pneumonia (Infections and infestations) | 8 (8) | 12 (12)
Urinary tract infection (Infections and infestations) | 19 (25) | 13 (17)
Alanine aminotransferase increased (Investigations) | 37 (53) | 43 (62)
Aspartate aminotransferase increased (Investigations) | 34 (43) | 38 (53)
Blood alkaline phosphatase increased (Investigations) | 23 (38) | 28 (32)
Blood bilirubin increased (Investigations) | 6 (18) | 12 (18)
Blood creatinine increased (Investigations) | 22 (32) | 17 (28)
Blood lactate dehydrogenase increased (Investigations) | 20 (35) | 14 (21)
Gamma-glutamyltransferase increased (Investigations) | 20 (25) | 14 (17)
Weight decreased (Investigations) | 21 (24) | 13 (17)
Decreased appetite (Metabolism and nutrition disorders) | 75 (93) | 44 (52)
Hyperglycaemia (Metabolism and nutrition disorders) | 22 (34) | 10 (15)
Hyperuricaemia (Metabolism and nutrition disorders) | 12 (19) | 7 (12)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 28 (53) | 12 (17)
Hypocalcaemia (Metabolism and nutrition disorders) | 17 (22) | 13 (21)
Hypokalaemia (Metabolism and nutrition disorders) | 22 (30) | 15 (25)
Hypomagnesaemia (Metabolism and nutrition disorders) | 38 (51) | 18 (28)
Hyponatraemia (Metabolism and nutrition disorders) | 41 (65) | 35 (59)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (26) | 20 (26)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (22) | 21 (23)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (15) | 12 (21)
Dizziness (Nervous system disorders) | 21 (24) | 17 (21)
Dysgeusia (Nervous system disorders) | 12 (15) | 13 (13)
Headache (Nervous system disorders) | 23 (27) | 18 (19)
Insomnia (Psychiatric disorders) | 24 (29) | 22 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (29) | 20 (22)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (27) | 26 (30)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 11 (14)
Alopecia (Skin and subcutaneous tissue disorders) | 88 (90) | 85 (86)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (16) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 48 (62) | 27 (32)
Rash (Skin and subcutaneous tissue disorders) | 52 (70) | 26 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT05224141/Prot_SAP_000.pdf